CLINICAL TRIAL: NCT00356512
Title: Physiologic Regulation of FGF-23
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060188; 06-D-0188
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-09-02

CONDITIONS: Hypoparathyroidism
Keywords: Phosphate; Vitamin D; Hypoparathyroidism; Phosphatonin; Clamp
MeSH Terms: conditions — Hypoparathyroidism

SUMMARY:
This study will explore the regulation of fibroblast growth factor-23 (FGF-23). It is a hormone recently identified as a regulator of the blood levels of phosphorus and vitamin D, both of which are essential for overall health and especially important for bone health. The parathyroid hormone (PTH) regulates phosphorus and calcium, but people with hypoparathyroidism or pseudohypoparathyroidism do not have sufficient PTH action. There are genetic diseases that influence FGF-23, causing abnormal metabolism of phosphorus and vitamin D, thus affecting the bones. Also, there are rare tumors that may cause overproduction of FGF-23 causing debilitating bone disease.

Patients ages 18 and older who have low PTH levels, or are resistant to PTH action, and take calcitriol and calcium supplements, who are not pregnant, and who do not have kidney disorders may be eligible for this study. During the 4-day study, patients will be provided with a controlled diet that has a lower than usual phosphorus content. On day 1, patients will be admitted to the NIH Clinic Center and undergo blood and urine tests to measure calcium, phosphorus, vitamin D, and FGF-23. They will continue with their regular medicine for hypoparathyroidism. On that day and throughout the study, patients will fast from 10:00 p.m. to 8:00 a.m. the following day. On day 2, patients will continue fasting until 4:00 p.m. A tube will be placed in the vein of each arm: one for drawing blood and the other for infusing calcium. Just one intravenous (IV) line will be used on the other days. Patients will receive calcium chloride for 8 hours, at a dose carefully monitored by a machine. The purpose is to bring the blood calcium level to the high normal range or just above. Blood and urine samples will be collected periodically, to check for effects of calcium chloride on FGF-23 and PTH. On days 3 and 4, patients will not take calcitriol and calcium but will receive injections of PTH, under the skin, two times each day. On day 3, blood and urine samples will be again be collected for analysis. On day 4, patients will receive one dose of calcitriol by IV. The total amount of blood drawn during this study will be about 5 ounces.

...

DETAILED DESCRIPTION:
Vitamin D and phosphate are central to normal mineral homeostasis and important in many physiologic functions including skeletal integrity. For several decades parathyroid hormone (PTH) has been recognized as a central regulator of serum vitamin D and phosphate levels. Recently, FGF-23 has been identified as central in the regulation of the metabolism of vitamin D and serum phosphorus. The organ primarily responsible for the physiologic production of FGF-23 appears to be the skeleton. The study of FGF-23 metabolism and its direct effect on mineral metabolism is confounded by the classic endocrine feedback loops that exist among serum calcium, phosphorus, 1,25-(OH)2-vitamin D (1,25-D), and PTH. It is possible that any of these (phosphorus, calcium, 1,25-D, and/or PTH) are important in the regulation of serum FGF-23. The goal of this study is to identify what factors regulate serum FGF-23.

To overcome the confounding effect of PTH, we will study patients deficient in PTH (hypoparathyroidism) or resistant to PTH at the kidney (pseudohypoparathyroidism type 1B, PHP1B). The kidney is one of the primary organs responsible for regulating serum phosphorus and generating 1,25-D. It is the target of PTH and FGF-23. While patients with PHP1B are resistant to the action of PTH at the kidney, they are sensitive to the action of PTH at the bone, the tissue that produces FGF-23. Physiologic manipulation of the serum phosphorus, 1,25-D, calcium, and PTH in subjects with hypoparathyroidism or PHP1B will allow for a nearly complete dissection of the factors that are potential regulators of serum FGF-23.

ELIGIBILITY:
* INCLUSION CRITERIA

Adult hypoparathyroid patients, as defined by low or inappropriately normal PTH levels despite hypocalcemia, who are on a stable treatment regimen of calcitriol and calcium supplementation, and who are willing to participate in the study will be eligible.

Adult PHP1B patients as defined by the clinical syndrome of elevated PTH and phosphorus and confirmed by methylation analysis of the GNAS gene.

EXCLUSION CRITERIA

Renal insufficiency as evidenced by a creatinine clearance of less than 50 ml/min

Medically unstable patients

Uncontrolled comorbid conditions, e.g., diabetes, coronary artery disease, congestive heart failure, or cerebrovascular disease.

Digitalis therapy

Patients on diuretic therapy, especially thiazides

Pregnant and lactating women

Patients whose hypoparathyroidism is caused by severe calcium-sensing receptor defects. These patients begin to have marked symptoms of "hypercalcemia" when the serum calcium is in the mid-normal range.

Patients under 18 years of age

Patients with history of any bone cancer, skeletal metastases or previous radiotherapy to the skeleton, unexplained elevations of serum alkaline phosphatase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-07-19; Primary Completion 2009-09-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kumar R. Phosphatonin--a new phosphaturetic hormone? (lessons from tumour-induced osteomalacia and X-linked hypophosphataemia). Nephrol Dial Transplant. 1997 Jan;12(1):11-3. doi: 10.1093/ndt/12.1.11. No abstract available. PMID 9027763
- [Background] Jonsson KB, Zahradnik R, Larsson T, White KE, Sugimoto T, Imanishi Y, Yamamoto T, Hampson G, Koshiyama H, Ljunggren O, Oba K, Yang IM, Miyauchi A, Econs MJ, Lavigne J, Juppner H. Fibroblast growth factor 23 in oncogenic osteomalacia and X-linked hypophosphatemia. N Engl J Med. 2003 Apr 24;348(17):1656-63. doi: 10.1056/NEJMoa020881. PMID 12711740
- [Background] Yamazaki Y, Okazaki R, Shibata M, Hasegawa Y, Satoh K, Tajima T, Takeuchi Y, Fujita T, Nakahara K, Yamashita T, Fukumoto S. Increased circulatory level of biologically active full-length FGF-23 in patients with hypophosphatemic rickets/osteomalacia. J Clin Endocrinol Metab. 2002 Nov;87(11):4957-60. doi: 10.1210/jc.2002-021105. PMID 12414858